CLINICAL TRIAL: NCT07053813
Title: Applying Population Management Best Practices to Preventive Genomic Medicine
Brief Title: Applying Population Management Best Practices to Preventative Genomic Medicine Trial
Acronym: CARE-HCS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Sarah Knerr, Assistant Professor, Health Systems and Population Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00021623; R01HG013021 (NIH)
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Neoplastic Syndromes, Hereditary
Keywords: hereditary cancer syndrome; pragmatic trial; population management; care coordination
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): No intervention
- Web resources (Experimental): Individuals randomized to web resources will be sent materials refined in Aim 1 (via patient portal and USPS mail) within 1-2 weeks after their birthday. Messages will be sent in English or preferred language noted in the EHR.
  Interventions: Behavioral: Web resources
- Personalized outreach (Experimental): Individuals randomized to personalized outreach will be contacted by the care coordinator in their birthday month for a brief phone call discussing due and overdue screening. The coordinator will attempt to contact patients up to 3 times to complete the phone conversation before considering them opting out of the intervention. If needed, the coordinator can place orders and pending referrals for PCP signature.
  Interventions: Behavioral: Personalized outreach

INTERVENTIONS:
Behavioral: Web resources — Mailed educational resources through portal and USPS mail
  Arms: Web resources
Behavioral: Personalized outreach — Phone call to discuss due and overdue screening and other personalized risk management recommendations
  Arms: Personalized outreach

SUMMARY:
Preventive genomic medicine, particularly identification of individuals with inherited cancer risk, can improve longevity and quality of life, yet adherence to risk management following cancer genomic testing is poor. The proposed research refines and evaluates two highly scalable population management interventions, web resources and personalized outreach, designed to improve access and use of recommended risk management following cancer genetic testing. Research activities will be conducted in a vertically integrated health system and federally qualified health center and will address post-testing quality and patient safety concerns that are minimizing patient benefit and slowing investments in real world genomic medicine implementation.

DETAILED DESCRIPTION:
Preventive genomic medicine, particularly identification of individuals with inherited cancer risk, provides health systems with the opportunity to improve longevity and quality of life for their patients. The ability to uncover substantially elevated risk of disease through genomic testing, act to reduce that risk, and improve outcomes while lowering costs has been the longstanding promise of genomic medicine. In the case of inherited cancer, however, adherence to recommended risk management following genomic testing is low. Further, our pilot data suggests that health systems are reluctant to expand cancer genomic testing without a clearer idea of how to manage tested patients over time. Our goal in this application is to address this roadblock to genomic medicine implementation. Specifically, we will demonstrate the benefits that adopting population management interventions following genomic testing can provide health systems, using hereditary cancer as a case example. We will revise and rigorously evaluate two population management interventions (web resources and personalized outreach) that improve timely patient outreach and end-to-end tracking without burdening providers. Web resources is a low-touch intervention that links patients with existing educational resources. Personalized outreach is a high-touch intervention that connects patients with a dedicated care manager to discuss risk management and provide care reminders.

Both interventions are highly scalable and mirror population management programs that health systems have used to support cancer screening, diabetes management, and other evidence-based care for decades. We will compare web resources and personalized outreach to usual care in a pragmatic hybrid type-1 randomized trial that engages patients captured in hereditary cancer registries within two health systems, Kaiser Permanente Northwest (KPNW) and Denver Health (DH). KPNW is a vertically integrated health system and DH is a federally qualified health center, providing two highly unique evaluation settings. Our primary effectiveness outcome is adherence to recommended cancer screening over one year. We will collect secondary implementation outcomes, including the acceptability, appropriateness, feasibility, sustainability, and costs of high- and low-touch intervention approaches. By providing clinical champions with essential data and tools to select and implement population management interventions that address critical gaps in post-testing quality and patient safety, this innovative project will advance preventive genomic medicine.

ELIGIBILITY:
Inclusion Criteria:

* Clinically actionable variant in at least one high penetrance cancer-related gene
* Age- and sex- eligible for guideline indicated risk management
* Remains eligible for risk management, given personal cancer and surgical history

Exclusion Criteria:

* Previously opted out of research
* Previously opted out of genetic research
* On hospice or palliative care
* Has advanced dementia or severe cognitive impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion time covered | 12 months following randomization
  Proportion time covered by recommended cancer screening

SECONDARY OUTCOMES:
Risk reducing surgery | 12 months following randomization
  Proportion completing one or more risk reducing surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Knerr, PhD, MPH, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Denver Health, Denver, Colorado
  - Kaiser Northwest, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
The University of Washington will create public use de-identified datasets of clinical trial data with an accompanying data dictionary, codes, and other documentation relevant to use.
Supporting Information: Study Protocol, SAP
Time Frame: IDP and supporting information will become available 6 months after the study's completion.
Access Criteria: The University of Washington will create Data Use Agreements with organizations that wish to access the dataset and accompanying documents.